CLINICAL TRIAL: NCT07046312
Title: Right Ventricular Strain in Detecting Subclinical Right Ventricular Systolic Dysfunction in Psoriatic Arthritis Patients: Relation to Serum Endostatin Level
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MD13/2025
Record Dates: First submitted 2025-05-19; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-05

CONDITIONS: Psoriatic Arthritis (PsA); Subclinical Right Ventricular Systolic Dysfunction
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: 30 control group matched as regards BMI, age and sex will be subjected to transthoracic echo and measuring serum endostatin level.
- Cases of Psoriatic arthritis patients: 30 PsA patients will be subjected to transthoracic echo, measuring serum endostatin level and modified composite psoriatic disease activity index

SUMMARY:
The aim is to assess early right ventricular systolic dysfunction in psoriatic arthritis patients using RV strain echocardiography

DETAILED DESCRIPTION:
Previous studies evaluated RV strain for detection of subclinical RV affection due to PAH in systemic lupus erythematosus. However , to our knowledge , the study of RV strain and its possible association with serum endostatin to detect subclinical right ventricular systolic dysfunction and its relation to PAH in PsA patient is still a novel. Our aim is to assess early right ventricular systolic dysfunction in psoriatic arthritis patients using RV strain Echocardiography.

To evaluate serum endostatin as an objective biomarker for Pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic arthritis patients according to CASPAR criteria
* Psoriatic arthritis patients without overt cardiovascular symptoms
* Patients with age between 20 to 50 years of age

Exclusion Criteria:

* Other systemic autoimmune diseases
* Patients with a history of known valvular disease, atrial fibrillation or any other arrhythmia , heart failure, ischemic cardiomyopathy severe obstructive pulmonary diseases and metabolic syndrome.
* Patients with medical disorders as renal, congenital heart diseases, hematological disorders and cancer patients.
* Patients taking certain drugs that have been confirmed to be risk factors for PAH such as appetite suppressant intake drugs (aminorex, fenfluramine derivatives and benfluorex) and chemotherapeutic agents.
* Family history of myocardial infarction, cerebrovascular disease or sudden death before the age of 65y in females and 55 y in males.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 patients with PsA and 30 matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Detecting subclinical right ventricular systolic dysfunction in PsA patients | Up to 24 months
  Detecting subclinical right ventricular systolic dysfunction in PsA using 2D strain transthoracic echo and its relation to serum endostatin level

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided